CLINICAL TRIAL: NCT02099110
Title: A Phase III, Randomized, Double-Blind, Multicenter Study to Evaluate the Efficacy and Safety of the Combination of Ertugliflozin (MK-8835/PF-04971729) With Sitagliptin Compared With Ertugliflozin Alone and Sitagliptin Alone, in the Treatment of Subjects With T2DM With Inadequate Glycemic Control on Metformin Monotherapy
Brief Title: Ertugliflozin and Sitagliptin Co-administration Factorial Study (VERTIS FACTORAL, MK-8835-005)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8835-005; MK-8835-005 (Other: Merck, Sharp & Dohme); B1521019 (Other: Pfizer); 2013-003698-82 (EudraCT Number)
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Results first posted 2017-11-01 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ertugliflozin; Sitagliptin Phosphate; Metformin; Insulin Glargine; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Ertugliflozin 5 mg + sitagliptin 100 mg (Experimental): Ertugliflozin 5 mg + sitagliptin 100 mg, oral, once daily for 52 weeks
  Interventions: Drug: Matching Placebo to Ertugliflozin 10 mg; Drug: Ertugliflozin 5 mg; Drug: Sitagliptin 100 mg; Drug: Metformin >= 1500 mg/day; Biological: Insulin Glargine Rescue Medication; Drug: Glimepiride Rescue Medication
- Ertugliflozin 15 mg + sitagliptin 100 mg (Experimental): Ertugliflozin 15 mg + sitagliptin 100 mg, oral, once daily for 52 weeks
  Interventions: Drug: Ertugliflozin 5 mg; Drug: Ertugliflozin 10 mg; Drug: Sitagliptin 100 mg; Drug: Metformin >= 1500 mg/day; Biological: Insulin Glargine Rescue Medication; Drug: Glimepiride Rescue Medication
- Ertugliflozin 5 mg (Experimental): Ertugliflozin 5 mg, oral, once daily for 52 weeks
  Interventions: Drug: Matching Placebo to Ertugliflozin 10 mg; Drug: Matching Placebo to sitagliptin 100 mg; Drug: Ertugliflozin 5 mg; Drug: Metformin >= 1500 mg/day; Biological: Insulin Glargine Rescue Medication; Drug: Glimepiride Rescue Medication
- Ertugliflozin 15 mg (Experimental): Ertugliflozin, oral, once daily for 52 weeks
  Interventions: Drug: Matching Placebo to sitagliptin 100 mg; Drug: Ertugliflozin 5 mg; Drug: Ertugliflozin 10 mg; Drug: Metformin >= 1500 mg/day; Biological: Insulin Glargine Rescue Medication; Drug: Glimepiride Rescue Medication
- Sitagliptin 100 mg (Active Comparator): Sitagliptin 100 mg, oral, once daily for 52 weeks
  Interventions: Drug: Matching Placebo to Ertugliflozin 5 mg; Drug: Matching Placebo to Ertugliflozin 10 mg; Drug: Sitagliptin 100 mg; Drug: Metformin >= 1500 mg/day; Biological: Insulin Glargine Rescue Medication; Drug: Glimepiride Rescue Medication

INTERVENTIONS:
Drug: Matching Placebo to Ertugliflozin 5 mg — Placebo to ertugliflozin 5 mg tablet, oral, once daily for 52 weeks during the double-blind treatment period
  Arms: Sitagliptin 100 mg
Drug: Matching Placebo to Ertugliflozin 10 mg — Placebo to ertugliflozin 10 mg tablet, oral, once daily for 52 weeks during the double-blind treatment period
  Arms: Ertugliflozin 5 mg; Ertugliflozin 5 mg + sitagliptin 100 mg; Sitagliptin 100 mg
Drug: Matching Placebo to sitagliptin 100 mg — Placebo to sitagliptin 100 mg tablet, oral, once daily for 52 weeks during the double-blind treatment period
  Arms: Ertugliflozin 15 mg; Ertugliflozin 5 mg
Drug: Ertugliflozin 5 mg — Ertugliflozin 5 mg tablet, oral, once daily for 52 weeks during the double-blind treatment period
  Other Names: MK-8835; PF-04971729
  Arms: Ertugliflozin 15 mg; Ertugliflozin 15 mg + sitagliptin 100 mg; Ertugliflozin 5 mg; Ertugliflozin 5 mg + sitagliptin 100 mg
Drug: Ertugliflozin 10 mg — Ertugliflozin 10 mg tablet, oral, once daily for 52 weeks during the double-blind treatment period
  Other Names: MK-8835; PF-04971729
  Arms: Ertugliflozin 15 mg; Ertugliflozin 15 mg + sitagliptin 100 mg
Drug: Sitagliptin 100 mg — Sitagliptin 100 mg tablet, oral, once daily for 52 weeks during the double-blind treatment period
  Other Names: JANUVIA®
  Arms: Ertugliflozin 15 mg + sitagliptin 100 mg; Ertugliflozin 5 mg + sitagliptin 100 mg; Sitagliptin 100 mg
Drug: Metformin >= 1500 mg/day — Metformin >= 1500 mg/day, tablets, oral, for 52 weeks while receiving blinded investigational product during the double-blind treatment period
  Other Names: Glucophage; Glucophage XR
Biological: Insulin Glargine Rescue Medication — Open-label insulin glargine, subcutaneous injection, as required as a rescue medication; dose determined per the investigator's discretion
  Other Names: Lantus
Drug: Glimepiride Rescue Medication — Open-label glimepiride tablets, oral, as required as a rescue medication, dose determined per the investigator's discretion
  Other Names: AMARYL

SUMMARY:
This is a study of co-administration of ertugliflozin (MK-8835/PF-04971729) and sitagliptin given together or alone along with metformin in participants with Type 2 diabetes mellitus (T2DM) and inadequate glycemic control on metformin monotherapy. The primary hypothesis of this study is that ertugliflozin 15 mg daily plus sitagliptin 100 mg daily provides greater hemoglobin A1C (A1C)-lowering compared with sitagliptin 100 mg daily alone.

DETAILED DESCRIPTION:
This study will include a 1-week screening period; an up to 12-week metformin titration/dose stabilization period; a 2-week single-blind placebo run-in period; a 52-week (26-week Phase A and 26-week Phase B) double-blind treatment period and a post-treatment telephone contact 14 days after the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus as per American Diabetes Association guidelines
* On metformin monotherapy (>=1500 mg/day) for >=8 weeks with a Visit 1/Screening A1C >=7.5% and <=11.0% (>=58 mmol/mol and <=97 mmol/mol) OR On metformin monotherapy (>=1500 mg/day) for <8 weeks with a Visit 1/Screening A1C >=7.5% and <=11.0% (>=58 mmol/mol and <=97 mmol/mol) OR On metformin monotherapy <1500 mg/day with a Visit 1/Screening A1C >=8.0% and <=11.5% (>=64 mmol/mol and <=102 mmol/mol)
* Body mass index (BMI) >=18.0 kg/m^2
* Male or female not of reproductive potential
* Female of reproductive potential who agrees to remain abstinent from heterosexual activity or to use 2 acceptable combinations of contraception

Exclusion Criteria:

* History of type 1 diabetes mellitus or ketoacidosis
* History of other specific types of diabetes (e.g., genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrinopathies, drug- or chemical-induced, and post-organ transplant
* A known hypersensitivity or intolerance to any sodium glucose co-transporter 2 (SGLT2) inhibitor or sitagliptin
* Has been treated with any of the following agents within 12 weeks of study start or during the pre-randomization period: Insulin of any type (except for short-term use [i.e., <=7 days] during concomitant illness or other stress), other injectable anti-hyperglycemic agents (e.g., pramlintide, exenatide, liraglutide), pioglitazone or rosiglitazone, other SGLT2 inhibitors, alpha glucosidase inhibitors or meglitinides, dipeptidyl-peptidase 4 inhibitor (DPP-4 inhibitor), sulfonylureas (SUs), bromocriptine (Cycloset™), colesevelam (Welchol™), any other antihyperglycemic agents (AHA) with the exception of the protocol-approved agents
* Is on a weight-loss program or weight-loss medication or other medication associated with weight changes and is not weight stable prior to study start
* Has undergone bariatric surgery within the past 12 months or >12 months and is not weight stable prior to study start
* A history of myocardial infarction, unstable angina, arterial revascularization, stroke, transient ischemic attack, or New York Heart Association (NYHA) functional class III-IV heart failure within 3 months of study start
* Active, obstructive uropathy or indwelling urinary catheter
* History of malignancy <=5 years prior to study start, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* A known history of human immunodeficiency virus (HIV)
* A blood dyscrasia or any disorder causing hemolysis or unstable red blood cells, or a clinically important hematological disorder (e.g. aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia)
* A medical history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease
* Any clinically significant malabsorption condition
* Current treatment for hyperthyroidism
* On thyroid replacement therapy and not on a stable dose for at least 6 weeks prior study start
* On a previous clinical study with ertugliflozin
* Estimated glomerular filtration rate (eGFR) (using the 4-variable Modification of Diet in Renal Disease Study Equation (MDRD) equation) <60 mL/min/1.73 m^2
* Serum creatinine >= 1.3 mg/dL (115 µmol/L) for males and >= 1.2 mg/dL (106 µmol/L) for females
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 times upper limit of normal
* Hemoglobin <12 g/dL (120 g/L) for males and <11 g/dL (110 g/L) for females.
* Participated in other studies involving investigational drug(s) 30 days prior to study start
* Surgical procedure within 6 weeks prior to study start or major surgery planned during the trial
* Positive urine pregnancy test
* Pregnant or breast-feeding, or planning to conceive during the trial, including 14 days following the last dose of study medication
* Planning to undergo hormonal therapy in preparation for egg donation during the trial, including 14 days following the last dose of study medication
* Routinely consumes >2 alcoholic drinks per day or >14 alcoholic drinks per week or engages in binge drinking
* Donated blood or blood products within 6 weeks of study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1233 (Actual)
Dates: Start 2014-04-22 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2016-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Pratley RE, Eldor R, Raji A, Golm G, Huyck SB, Qiu Y, Sunga S, Johnson J, Terra SG, Mancuso JP, Engel SS, Lauring B. Ertugliflozin plus sitagliptin versus either individual agent over 52 weeks in patients with type 2 diabetes mellitus inadequately controlled with metformin: The VERTIS FACTORIAL randomized trial. Diabetes Obes Metab. 2018 May;20(5):1111-1120. doi: 10.1111/dom.13194. Epub 2018 Jan 25. PMID 29266675
- [Derived] Fediuk DJ, Sahasrabudhe V, Dawra VK, Zhou S, Sweeney K. Population Pharmacokinetic Analyses of Ertugliflozin in Select Ethnic Populations. Clin Pharmacol Drug Dev. 2021 Nov;10(11):1297-1306. doi: 10.1002/cpdd.970. Epub 2021 Jul 2. PMID 34213819
- [Derived] Gallo S, Raji A, Calle RA, Pong A, Meyer C. The effects of ertugliflozin on beta-cell function: Pooled analysis from four phase 3 randomized controlled studies. Diabetes Obes Metab. 2020 Dec;22(12):2267-2275. doi: 10.1111/dom.14149. Epub 2020 Aug 27. PMID 32700393
- [Derived] Gallo S, Calle RA, Terra SG, Pong A, Tarasenko L, Raji A. Effects of Ertugliflozin on Liver Enzymes in Patients with Type 2 Diabetes: A Post-Hoc Pooled Analysis of Phase 3 Trials. Diabetes Ther. 2020 Aug;11(8):1849-1860. doi: 10.1007/s13300-020-00867-1. Epub 2020 Jul 9. PMID 32648108
- [Derived] Patel S, Hickman A, Frederich R, Johnson S, Huyck S, Mancuso JP, Gantz I, Terra SG. Safety of Ertugliflozin in Patients with Type 2 Diabetes Mellitus: Pooled Analysis of Seven Phase 3 Randomized Controlled Trials. Diabetes Ther. 2020 Jun;11(6):1347-1367. doi: 10.1007/s13300-020-00803-3. Epub 2020 May 5. PMID 32372382
- [Derived] Liu J, Tarasenko L, Pong A, Huyck S, Wu L, Patel S, Hickman A, Mancuso JP, Gantz I, Terra SG. Efficacy and safety of ertugliflozin across racial groups in patients with type 2 diabetes mellitus. Curr Med Res Opin. 2020 Aug;36(8):1277-1284. doi: 10.1080/03007995.2020.1760228. Epub 2020 May 13. PMID 32324082
- [Derived] Liu J, Tarasenko L, Pong A, Huyck S, Patel S, Hickman A, Mancuso JP, Ellison MC, Gantz I, Terra SG. Efficacy and safety of ertugliflozin in Hispanic/Latino patients with type 2 diabetes mellitus. Curr Med Res Opin. 2020 Jul;36(7):1097-1106. doi: 10.1080/03007995.2020.1760227. Epub 2020 May 13. PMID 32324065
- [Derived] Liu J, Patel S, Cater NB, Wu L, Huyck S, Terra SG, Hickman A, Darekar A, Pong A, Gantz I. Efficacy and safety of ertugliflozin in East/Southeast Asian patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2020 Apr;22(4):574-582. doi: 10.1111/dom.13931. Epub 2020 Jan 3. PMID 31797522

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 21 countries and included 242 trial centers.
Pre-assignment Details: Participants on ≥1500 mg/day of metformin for ≥8 weeks with A1C ≥7.5 and ≤11% at screening could directly enter a 2-week, single-blind, placebo run-in period. Participants who did not meet these criteria, received diet/exercise counseling and metformin titration (as necessary) for ~8 weeks before entering the 2-week, placebo run-in period.
Period: Overall Study
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Sitagliptin 100 mg | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg
Started | 250 | 248 | 247 | 243 | 245
Treated | 250 | 248 | 247 | 243 | 244
Completed | 226 | 217 | 219 | 221 | 218
Not Completed | 24 | 31 | 28 | 22 | 27
Not completed — Protocol Violation | 2 | 1 | 0 | 3 | 1
Not completed — Participant moved | 1 | 1 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 7 | 11 | 13 | 9 | 13
Not completed — Adverse Event | 3 | 5 | 2 | 3 | 2
Not completed — Lost to Follow-up | 6 | 12 | 11 | 5 | 6
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Screen failure | 0 | 0 | 0 | 0 | 1
Not completed — Non-compliance with study drug | 2 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 3 | 0 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population was the All-Participants-As-Treated population. One participant randomized to the Ertugliflozin 15 mg + Sitagliptin 100 mg arm did not receive study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Sitagliptin 100 mg | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg | Total
Number analyzed (Participants) | 250 | 248 | 247 | 243 | 244 | 1232
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.1 (10.1) | 55.3 (9.5) | 54.8 (10.7) | 55.2 (10.4) | 55.1 (9.8) | 55.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 114 | 93 | 120 | 118 | 568
  Male | 127 | 134 | 154 | 123 | 126 | 664
Baseline Hemoglobin A1C (A1C) [Mean (Standard Deviation); unit: Percent] — A1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). Population: Participants with baseline data for A1C.
  Percent
    number analyzed (Participants) | 244 | 247 | 242 | 237 | 241 | 1211
    (all) | 8.6 (1.0) | 8.6 (1.0) | 8.5 (1.0) | 8.6 (1.0) | 8.6 (1.0) | 8.6 (1.0)
Baseline Body Weight [Mean (Standard Deviation); unit: Kilograms] | 88.6 (22.2) | 88.0 (20.3) | 89.8 (23.4) | 89.5 (20.8) | 87.5 (20.5) | 88.7 (21.5)
Baseline Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] — Blood glucose was measured on a fasting basis after at least a 10-hour fast. Population: Participants with baseline data for Fasting Plasma Glucose.
  mg/dL
    number analyzed (Participants) | 250 | 247 | 246 | 240 | 241 | 1224
    (all) | 184.1 (52.2) | 179.5 (45.7) | 177.4 (46.6) | 183.8 (44.3) | 177.2 (49.4) | 180.4 (47.8)
Static Beta-Cell Sensitivity to Glucose Index [Mean (Standard Deviation); unit: SBCSGI (10^-9min^-1)] — Static beta-cell sensitivity to glucose index (SBCSGI) estimates the ratio of insulin secretion (expressed in pmol/min) related to above-basal glucose concentration (expressed in mmol/L * L) following a meal. Blood samples were collected before and after a standard meal and glucose, insulin, and C-peptide levels were analyzed. The C-peptides minimal model was used to estimate the insulin secretion rate. Analysis was performed with non-linear least squares using the Software Architecture Analysis Method (SAAM) II software. SBCSGI was expressed in units of 10^-9 min^-1. Population: Participants with baseline data for SBCSGI.
  SBCSGI (10^-9min^-1)
    number analyzed (Participants) | 58 | 58 | 55 | 48 | 50 | 269
    (all) | 20.9 (26.1) | 18.0 (16.3) | 20.2 (21.2) | 20.0 (16.6) | 19.3 (21.0) | 19.7 (20.5)
Sitting Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 129.7 (12.5) | 128.9 (12.5) | 128.3 (12.2) | 130.2 (12.6) | 129.1 (13.3) | 129.3 (12.6)
Baseline estimated glomerular filtration rate, eGFR [Mean (Standard Deviation); unit: mL/min/1.73m^2] — eGFR is a parameter used to assess kidney function. Population: Participants with baseline data for eGFR.
  mL/min/1.73m^2
    number analyzed (Participants) | 250 | 248 | 247 | 242 | 244 | 1231
    (all) | 91.9 (20.6) | 92.8 (21.4) | 92.6 (18.2) | 91.9 (20.4) | 92.6 (19.2) | 92.4 (20.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C at Week 26: Excluding Rescue Approach
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). This change from baseline reflects the Week 26 A1C minus the Week 0 A1C. Excluding recue approach data analysis excluded all data following the initiation of rescue therapy at any time point, in order to avoid the confounding influence of the rescue therapy.
Time Frame: Baseline and Week 26
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment, had a baseline measurement or a post-randomization measurement for the A1C change from baseline at Week 26 analysis endpoint subsequent to at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Sitagliptin 100 mg | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg
Number analyzed (Participants) | 250 | 248 | 247 | 243 | 244
Percentage | -1.02 [-1.14 to -0.90] | -1.08 [-1.20 to -0.96] | -1.05 [-1.17 to -0.93] | -1.49 [-1.61 to -1.36] | -1.52 [-1.64 to -1.40]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Ertugliflozin 5 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis — Constrained longitudinal data analysis (cLDA) model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment. Time was treated as a categorical variable; Difference in the least squares means = -0.46, 95% CI 2-sided [-0.63 to -0.30]
Statistical Analysis 2: Comparison: Sitagliptin 100 mg vs Ertugliflozin 5 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis — cLDA model with fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment. Time was treated as a categorical variable; Difference in the least squares means = -0.43, 95% CI 2-sided [-0.60 to -0.27]
Statistical Analysis 3: Comparison: Ertugliflozin 15 mg vs Ertugliflozin 15 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 2]; Difference in the least squares means = -0.44, 95% CI 2-sided [-0.61 to -0.27]
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Ertugliflozin 15 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 2]; Difference in the least squares means = -0.47, 95% CI 2-sided [-0.63 to -0.30]

2. Primary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE): Including Rescue Approach
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. Including rescue approach data analysis included data following the initiation of rescue therapy.
Time Frame: Up to 54 weeks
Population: The analysis population consists of all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Sitagliptin 100 mg | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg
Number analyzed (Participants) | 250 | 248 | 247 | 243 | 244
Percentage of participants | 62.0 | 57.7 | 57.5 | 58.8 | 55.7
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Ertugliflozin 5 mg + Sitagliptin 100 mg; Test type: Superiority or Other; Difference in % vs Ertugliflozin 5 mg = -3.2, 95% CI 2-sided [-11.7 to 5.5] — Based on Miettinen & Nurminen method
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Ertugliflozin 15 mg + Sitagliptin 100 mg; Test type: Superiority or Other; Difference in % vs. Ertugliflozin 15 mg = -1.9, 95% CI 2-sided [-10.6 to 6.8] — Based on Miettinen & Nurminen method
Statistical Analysis 3: Comparison: Sitagliptin 100 mg vs Ertugliflozin 5 mg + Sitagliptin 100 mg; Test type: Superiority or Other; Difference in % vs. Sitagliptin 100 mg = 1.4, 95% CI 2-sided [-7.4 to 10.1] — Based on Miettinen & Nurminen method
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Ertugliflozin 15 mg + Sitagliptin 100 mg; Test type: Superiority or Other; Difference in % vs. Sitagliptin 100 mg = -1.8, 95% CI 2-sided [-10.5 to 7.0] — Based on Miettinen & Nurminen method

3. Primary Outcome: Percentage of Participants Who Discontinued Study Treatment Due to an AE: Including Rescue Approach
Description: as for outcome 2
Time Frame: Up to 52 weeks
Population: The analysis population consists of all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Sitagliptin 100 mg | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg
Number analyzed (Participants) | 250 | 248 | 247 | 243 | 244
Percentage of participants | 3.2 | 3.2 | 2.8 | 3.3 | 3.7
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Ertugliflozin 5 mg + Sitagliptin 100 mg; Test type: Superiority or Other; Difference in % vs. Ertugliflozin 5 mg = 0.1, 95% CI 2-sided [-3.3 to 3.6] — Based on Miettinen & Nurminen method
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Ertugliflozin 15 mg + Sitagliptin 100 mg; Test type: Superiority or Other; Difference in % vs. Ertugliflozin 15 mg = 0.5, 95% CI 2-sided [-3.0 to 4.0] — Based on Miettinen & Nurminen method
Statistical Analysis 3: Comparison: Sitagliptin 100 mg vs Ertugliflozin 5 mg + Sitagliptin 100 mg; Test type: Superiority or Other; Difference in % vs. Sitagliptin 100 mg = 0.5, 95% CI 2-sided [-2.9 to 3.9] — Based on Miettinen & Nurminen method
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Ertugliflozin 15 mg + Sitagliptin 100 mg; Test type: Superiority or Other; Difference in % vs. Sitagliptin 100 mg = 0.9, 95% CI 2-sided [-2.5 to 4.4] — Based on Miettinen & Nurminen method

4. Secondary Outcome: Change From Baseline in Body Weight at Week 26: Excluding Rescue Approach
Description: This change from baseline reflects the Week 26 body weight minus the Week 0 body weight. Excluding recue approach data analysis excluded all data following the initiation of rescue therapy at any time point, in order to avoid the confounding influence of the rescue therapy.
Time Frame: Baseline and Week 26
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment, had a baseline measurement or a post-randomization measurement for the body weight change from baseline at Week 26 analysis endpoint subsequent to at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Sitagliptin 100 mg | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg
Number analyzed (Participants) | 250 | 248 | 247 | 243 | 244
Kilograms | -2.69 [-3.13 to -2.25] | -3.74 [-4.18 to -3.29] | -0.67 [-1.12 to -0.22] | -2.52 [-2.97 to -2.07] | -2.94 [-3.39 to -2.49]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Ertugliflozin 5 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis — cLDA model including fixed effects for treatment, time, baseline eGFR (continuous) and the interaction of time by treatment. Time was treated as a categorical variable; Difference in the least squares means = -1.85, 95% CI 2-sided [-2.48 to -1.22]
Statistical Analysis 2: Comparison: Sitagliptin 100 mg vs Ertugliflozin 15 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, Constrained logitudinal data analysis — [p-value comment as in outcome 4, analysis 1]; Difference in the least squares means = -2.27, 95% CI 2-sided [-2.90 to -1.64]

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 26 - Excluding Rescue Approach
Description: Blood glucose was measured on a fasting basis after at least a 10-hour fast. This change from baseline reflects the Week 26 FPG minus the Week 0 FPG. Excluding recue approach data analysis excluded all data following the initiation of rescue therapy at any time point, in order to avoid the confounding influence of the rescue therapy.
Time Frame: Baseline and Week 26
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment, had a baseline measurement or a post-randomization measurement for the FPG change from baseline at Week 26 analysis endpoint subsequent to at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Sitagliptin 100 mg | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg
Number analyzed (Participants) | 250 | 248 | 247 | 243 | 244
mg/dL | -35.73 [-40.04 to -31.42] | -36.91 [-41.21 to -32.62] | -25.56 [-29.93 to -21.19] | -43.96 [-48.29 to -39.63] | -48.70 [-53.01 to -44.39]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Ertugliflozin 5 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.004, cLDA — [p-value comment as in outcome 4, analysis 1]; Difference in the least squares means = -8.23, 95% CI 2-sided [-13.82 to -2.65]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Ertugliflozin 15 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, cLDA — [p-value comment as in outcome 4, analysis 1]; Difference in the least squares means = -11.79, 95% CI 2-sided [-17.35 to -6.23]
Statistical Analysis 3: Comparison: Sitagliptin 100 mg vs Ertugliflozin 5 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, cLDA — [p-value comment as in outcome 4, analysis 1]; Difference in the least squares means = -18.40, 95% CI 2-sided [-24.03 to -12.77]
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Ertugliflozin 15 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, cLDA — [p-value comment as in outcome 4, analysis 1]; Difference in the least squares means = -23.14, 95% CI 2-sided [-28.76 to -17.53]

6. Secondary Outcome: Percentage of Participants Achieving a Hemoglobin A1C of <7% (<53 mmol/Mol) (Raw Proportions): Excluding Rescue Approach
Description: A1C is blood marker used to report average blood glucose levels over a prolonged periods of time and is reported as a percentage (%). Excluding recue approach data analysis excluded all data following the initiation of rescue therapy at any time point, in order to avoid the confounding influence of the rescue therapy.
Time Frame: Week 26
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment, had a post-randomization measurement for the A1C change from baseline at Week 26 analysis endpoint subsequent to at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Sitagliptin 100 mg | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg
Number analyzed (Participants) | 250 | 248 | 247 | 243 | 244
Percentage of participants | 26.4 | 31.9 | 32.8 | 52.3 | 49.2
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Ertugliflozin 5 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Adjusted Odds Ratio using a logistic regression model fitted with fixed effects for treatment, covariates for baseline A1C and baseline eGFR; Odds Ratio (OR) = 4.14, 95% CI 2-sided [2.68 to 6.40]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Ertugliflozin 15 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; Odds Ratio (OR) = 2.53, 95% CI 2-sided [1.68 to 3.83]
Statistical Analysis 3: Comparison: Sitagliptin 100 mg vs Ertugliflozin 5 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]; Odds Ratio (OR) = 2.95, 95% CI 2-sided [1.92 to 4.54]
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Ertugliflozin 15 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Adjusted Odds Ratio using a logistic regression model fitted with fixed effects for treatment, covariates for baseline A1C and baseline eGFR; Odds Ratio (OR) = 2.56, 95% CI 2-sided [1.69 to 3.89]

7. Secondary Outcome: Change From Baseline in Static Beta-Cell Sensitivity to Glucose Index at Week 26; Excluding Rescue Approach
Description: Static beta-cell sensitivity to glucose index (SBCSGI) estimates the ratio of insulin secretion (expressed in pmol/min) related to above-basal glucose concentration (expressed in mmol/L * L) following a meal. Blood samples were collected before and after a standard meal and glucose, insulin, and C-peptide levels were analyzed. The C-peptides minimal model was used to estimate the insulin secretion rate (ISR). Analysis included both non-model-based [including insulinogenic index with C-peptide, glucose area under the curve (AUC)/insulin AUC] and model-based [beta cell function and insulin secretion rate at 9 mM glucose] testing. Analysis was performed with non-linear least squares using the Software Architecture Analysis Method (SAAM) II software. SBCSGI was expressed in units of 10^-9 min^-1. Excluding rescue approach data analysis excluded all data following the initiation of rescue therapy at any time point, in order to avoid the confounding influence of the rescue therapy.
Time Frame: 30 min. before and 0, 15, 30, 60, 90, 120, and 180 minutes following the start of the standard meal at Baseline and Week 26
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment, had a baseline measurement or a post-randomization measurement for the beta-cell responsivity static component change from baseline at Week 26 analysis endpoint subsequent to at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: SBCSGI (10^-9min^-1)
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Sitagliptin 100 mg | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg
Number analyzed (Participants) | 66 | 67 | 63 | 55 | 61
SBCSGI (10^-9min^-1) | 8.62 [1.28 to 15.96] | 9.71 [2.29 to 17.13] | 21.11 [13.55 to 28.67] | 16.24 [8.36 to 24.11] | 11.51 [3.76 to 19.26]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Ertugliflozin 5 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.155, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 2]; Difference in the least squares means = 7.61, 95% CI 2-sided [-2.90 to 18.13]
Statistical Analysis 2: Comparison: Sitagliptin 100 mg vs Ertugliflozin 5 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.369, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 2]; Difference in the least squares means = -4.87, 95% CI 2-sided [-15.54 to 5.80]
Statistical Analysis 3: Comparison: Ertugliflozin 15 mg vs Ertugliflozin 15 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.734, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 2]; Difference in the least squares means = 1.81, 95% CI 2-sided [-8.66 to 12.27]
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Ertugliflozin 15 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.075, Difference in the least squares means — [p-value comment as in outcome 1, analysis 2]; Difference in the least squares means = -9.59, 95% CI 2-sided [-20.17 to 0.98]

8. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure at Week 26: Excluding Rescue Approach
Description: This change from baseline reflects the Week 26 systolic blood pressure minus the Week 0 systolic blood pressure. Excluding recue approach data analysis excluded all data following the initiation of rescue therapy at any time point, in order to avoid the confounding influence of the rescue therapy.
Time Frame: Baseline and Week 26
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment, had a baseline measurement or a post-randomization measurement for the systolic blood pressure change from baseline at Week 26 analysis endpoint subsequent to at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Sitagliptin 100 mg | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg
Number analyzed (Participants) | 250 | 248 | 247 | 243 | 245
mm Hg | -3.89 [-5.28 to -2.50] | -3.69 [-5.08 to -2.30] | -0.66 [-2.07 to 0.76] | -3.42 [-4.82 to -2.03] | -3.67 [-5.06 to -2.29]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Ertugliflozin 5 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.005, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 2]; Difference in the least squares means = -2.76, 95% CI 2-sided [-4.69 to -0.83]
Statistical Analysis 2: Comparison: Sitagliptin 100 mg vs Ertugliflozin 15 mg + Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.002, Constrained longitudinal data analysis — [p-value comment as in outcome 1, analysis 2]; Difference in the least squares means = -3.01, 95% CI 2-sided [-4.94 to -1.09]

ADVERSE EVENTS:
Time Frame: Up to 54 weeks
Description: The safety population consisted of all randomized participants who took at least one dose of trial treatment. Participants were included in the treatment group corresponding to the trial treatment they actually took. This analysis included events that occurred following the initiation of rescue therapy.
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Sitagliptin 100 mg | Ertugliflozin 5 mg + Sitagliptin 100 mg | Ertugliflozin 15 mg + Sitagliptin 100 mg
Serious Adverse Events (participants affected / at risk) | 12/250 | 5/248 | 8/247 | 9/243 | 12/244
Other Adverse Events (participants affected / at risk) | 36/250 | 43/248 | 28/247 | 31/243 | 38/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertugliflozin 5 mg (N=250) | Ertugliflozin 15 mg (N=248) | Sitagliptin 100 mg (N=247) | Ertugliflozin 5 mg + Sitagliptin 100 mg (N=243) | Ertugliflozin 15 mg + Sitagliptin 100 mg (N=244)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Microvascular coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femoral hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis orbital (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodal marginal zone B-cell lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertugliflozin 5 mg (N=250) | Ertugliflozin 15 mg (N=248) | Sitagliptin 100 mg (N=247) | Ertugliflozin 5 mg + Sitagliptin 100 mg (N=243) | Ertugliflozin 15 mg + Sitagliptin 100 mg (N=244)
Hypoglycaemia (Metabolism and nutrition disorders) | 12 (25) | 13 (29) | 11 (22) | 9 (17) | 20 (42)
Nasopharyngitis (Infections and infestations) | 6 (6) | 13 (14) | 6 (7) | 12 (14) | 12 (13)
Urinary tract infection (Infections and infestations) | 20 (24) | 19 (23) | 13 (13) | 14 (18) | 8 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.